CLINICAL TRIAL: NCT00343759
Title: Presurgical Therapy With Lapatinib to Explore Molecular Determinants of Response to EGFR/erbB2 Targeted Therapy
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 803893; UPCC 12104
Record Dates: First submitted 2006-06-21; First posted 2006-06-23 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Breast Cancer
Keywords: Breast cancer; Tyrosine kinase inhibitors; Lapatinib; Biologic response modifiers; Magnetic resonance imaging; Treatment-naive, operable
MeSH Terms: conditions — Breast Neoplasms | interventions — Lapatinib

INTERVENTIONS:
Drug: Lapatinib — Patients will take 14 days of Lapatinib prior to definitive surgery.

SUMMARY:
The purpose of this study is to see what kinds of breast tumors will respond to lapatinib. Lapatinib is an experimental medicine which may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically-confirmed by either core or fine needle biopsy primary invasive carcinoma of the breast;
* AJCC T2-T3 disease (>2.0 cm without chest wall or skin invasion) by at least one imaging modality (either mammogram, ultrasound, or MRI) - entry criteria is based on radiologic staging and not final pathologic staging;
* ECOG performance status 0-1 (Karnofsky ≥ 70%
* Any lymph node status, hormone receptor status, and level of erbB2 expression
* No prior chemotherapy, hormonal therapy or radiation therapy to the affected breast for current or previous malignancy;
* Cardiac ejection fraction >50% or within the institutional range of normal;
* Patients must have normal organ and marrow function defined as: Leukocyte count >3000/uL; Absolute neutrophil count (ANC) ≥ 1,500/mm3, platelets > 100,000/mm3, and hemoglobin ≥ 8 gm/dl; Serum creatinine ≤ 1.5 times ULN, or 24-hour creatinine clearance ≥ 75 cc/min; Serum bilirubin ≤ 1.5 times ULN; SGOT ≤ 2.5 times ULN; alkaline phosphatase ≤ 2.5 ULN times ULN.
* The effects of lapatinib on the developing human fetus at the recommended therapeutic dose are unknown. For this reason, women of child-bearing potential and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she must inform her treating physician immediately.
* Ability to understand and the willingness to sign written informed consent document.

Exclusion Criteria:

* AJCC T1, T4, or stage 4 disease;
* Patients may not have undergone incisional or excisional biopsy of their tumor;
* Patients may not be receiving any other investigational agents;
* Absolute contraindication to MRI imaging (cardiac pacemaker or any non-removable metallic foreign object in the body);
* On chronic therapy with any known inducer or inhibitor of CYP3A4
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant or lactating women are excluded from this study because lapatinib is a tyrosine kinase inhibitor with the potential for teratogenic or abortifacient effects.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2006-06; Primary Completion 2009-05 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Change in downstream effector levels in biologic responders to lapatinib as determined by degree of change in proliferation and apoptosis compared to biologic non-responders. | Study completion

SECONDARY OUTCOMES:
To describe the biologic response rate, defined by induction of apoptosis, to Lapatinib in a pre-surgical, treatment-naïve breast cancer population. | Study completion

CONTACTS AND LOCATIONS:
Overall Officials: Angela DeMichele, M.D., Principal Investigator — University of Pennsylvania
Locations (1):
- Abramson Cancer Center of University of Pennsylvania, Philadelphia, Pennsylvania, United States